CLINICAL TRIAL: NCT03371524
Title: A Prospective RegistrY of Cardiac Echographic Loops
Acronym: ARYEL
Status: Completed | Type: Observational
Sponsor: Cardiawave SA (Industry)
Responsible Party: Sponsor
Other Study IDs: ARYEL
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Calcified Aortic Valve
MeSH Terms: conditions — Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Native valves_30 seconds loops: Patient with calcified aortic stenosis on native valve: record of a 30 second loop during routine cardiac echography.
  Interventions: Other: Cardiac Echography
- Native valves_30 and 60 seconds loops: Patient with calcified aortic stenosis on native valve: record of a 30 second loop and a 60 second loop during routine cardiac echography.
  Interventions: Other: Cardiac Echography
- Bioprosthesis_30 seconds loops: Patient with calcified aortic stenosis on bioprosthesis: record of a 30 second loop during routine cardiac echography.
  Interventions: Other: Cardiac Echography

INTERVENTIONS:
Other: Cardiac Echography — While routine cardiac echography is performed on patients with calcified aortic valve, a 30 second loop is recorded.

SUMMARY:
CARDIAWAVE, a French start-up founded in 2014, aims to develop a new non-invasive therapy to treat patients suffering from Aortic Valve Stenosis (AS) who are not candidates to validated treatment of AS, i.e. TAVI (Transcatheter Aortic Valve Implantation) or SAVR (Surgical Aortic Valve Replacement). This therapy consists in focusing ultrasound on aortic valve transthoracically and use high energy to soften calcification from the target valve. In order to do so, we develop a device able to deliver high energy ultrasounds to a targeted valve thanks to the synchronization of patient hearts live imaging and therapy in real time.

Live imaging will use an algorithm to realize 'valve tracking': an automatic detection of aortic valve position and shape as fast as image acquisition time. In order to develop and validate this 'valve tracking' algorithm, CARDIAWAVE requires cardiac echographic loops of patients with aortic valve calcification, with 30 seconds or 60 seconds recording.

The objective of the present study is to develop and validate the 'valve tracking' processing algorithm of CARDIAWAVE.

ARYEL is a prospective, multicenter, non-interventional study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 y.o
* Patients with a confirmed diagnosis of Aortic valve calcification on native valve or bioprosthesis
* Patients with planned cardiac transthoracic echography for 'Aortic valve calcification' follow-up
* Patients who have signed Informed Consent Form
* Patients affiliated to French social security or equivalent

Exclusion Criteria:

* Patients allergic to echographic gel
* Patients with "hostile thorax": serious cutaneous irradiation injury or major thoracic deformity.
* Low echogenicity
* Patients with mild or high abundance pericardic effusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed calcified aortic stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Validation of the 'valve tracking' processing algorithm of CARDIAWAVE. | Through study completion, up to 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Caen, Caen
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Charles Nicolle, Rouen

IPD SHARING:
Plan to Share IPD: No